CLINICAL TRIAL: NCT06895629
Title: Feasibility and Efficacy of PRO-MAMA - a Novel Occupational Therapy Intervention for Promoting Participation, Health and Wellbeing Among Older Mothers After Stroke and Other Chronic Conditions.
Brief Title: Feasibility and Efficacy of PRO-MAMAS
Acronym: PRO-MAMAS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Debbie Rand, Professor Debbie Rand, Tel Aviv University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-MAMAS 0010055-1
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-05

CONDITIONS: Chronic Stroke
MeSH Terms: interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRO-MAMAS (Experimental): All participants will receive PRO-MAMAS - a novel occupational therapy intervention.
  PRO-MAMAS will include 8 sessions (2 sessions per week for 4 weeks). PRO-MAMAS will include small group of 5-8 participants, so approximately 4 rounds of PRO-MAMAS will be needed to reach 30 participants
  Interventions: Behavioral: PRO-MAMAS (Promoting participation, health and wellbeing through meaningful maternal-role activities after stroke and other chronic conditions)

INTERVENTIONS:
Behavioral: PRO-MAMAS (Promoting participation, health and wellbeing through meaningful maternal-role activities after stroke and other chronic conditions) — PRO-MAMAS - a novel occupational therapy intervention program to promote participation, health and wellbeing of older mothers with chronic stroke and other chronic conditions.

SUMMARY:
This experimental design will assess the feasibility & initial effectiveness of PRO-MAMAS (promoting participation, health and wellbeing through meaningful maternal-role activities after stroke and other chronic conditions) - a novel occupational therapy intervention program to promote participation, health and wellbeing of older mothers with chronic stroke.

Assessments will be conducted at three time points: baseline, pre, post the Pro-MAMA intervention

DETAILED DESCRIPTION:
This study aims to test the feasibility and initial effectiveness of PRO-MAMAS (promoting participation, health and wellbeing through meaningful maternal-role activities after stroke and other chronic conditions) in improving participation, health and wellbeing among older community dwelling mothers with chronic stroke and other chronic conditions.

PRO-MAMAS is a group intervention that aims to promote the health and wellbeing of older mothers with chronic stroke and other chronic conditions by using meaningful maternal-role activities as a motivational mean for participation. The intervention will include group discussions and practice, analysis of facilitators and barriers for participation, and home exercise. PRO-MAMAS will focus on raising awareness to meaningful maternal-role activities, identifying facilitators and barriers for participation and problem solving to enhance meaningful participation.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Aged 70 and older
* Mothers (have at least one live and healthy child)
* With chronic stroke (at lease six months from stroke onset) or other age-related chronic conditions
* That live at home
* That they can walk independently (with or without a walking aid)
* Without significant cognitive decline (MoCA ≥19)

Ages: 70 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with PRO-MAMAS intervention | Post intervention (week 8)
  A self-report questionnaire assessing the satisfaction with the novel intervention. The participants rate their agreement with statements relating to the intervention on a scale of 1=not at all to 5=very much.
Change in scores of the Canadian Occupational Performance Measure (COPM) | Change from pre (week 3) to post intervention (week 8)
  Change in scores of performance and satisfaction of performance for therapeutic goals that the participants define as important to them. Goals will focus on maternal-role and general participation.
Change in scores of the Short Form Health Survey (SF-12) | Change from pre (week 3) to post intervention (week 8)
  The SF-12 is a 12-question assessment measuring physical and mental health, including areas such as physical functioning, pain, social functioning, and emotional well-being. It generates Physical (PCS) and Mental (MCS) Component Summary scores, ranging from 0 to 100, with higher scores indicating better health.
Change in scores of the Satisfaction with Life Scale (SWLS) | Change from pre (week 3) to post intervention (week 8)
  SWLS is a 5-item questionnaire that measures overall life satisfaction. Respondents rate their agreement with statements on a 7-point scale (1 = strongly disagree, 7 = strongly agree), producing a total score ranging from 5 to 35, with higher scores indicating greater life satisfaction.

SECONDARY OUTCOMES:
Change in the Older adults' - Meaningful Maternal-role Activities Assessment (O-MAMA) | Change from baseline (week 0) to post intervention (week 8)
  A self-report questionnaire, includes 37 items and measures participation of older mothers in meaningful maternal-role activities, producing two total scores: percent-Participation and percent-Non-Participation. Higher percent-Participation scores indicate more participation in meaningful maternal-role activities whereas higher percent-Non-Participation scores indicate less participation in these activities.
Change in Reintegration to Normal Living Index (RNL) | Change from baseline (week 0) to post intervention (week 8)
  A self-reported questionnaire for assessing participation in various contexts such as recreational activity and family roles. Scores range between 10-100, higher scores indicate more participation.
The Lawton Instrumental Activities of Daily Living (IADLq) | Change from pre (week 0) to post intervention (week 8)
  A self-report questionnaire, assesses independence in tasks such as shopping. Scores range between 0-23 points, higher scores indicate more independence.
Change in Timed Up and Go (TUG) | Change from pre (week 3) to post intervention (week 8)
  An assessment of mobility, measures the time (in seconds) it takes for an individual to stand up from a chair, walk 3 meters, turn, walk back, and sit down. A longer completion time indicates reduced mobility and a higher fall risk.
Change in ABILHAND | Change from pre (week 3) to post intervention (week 8)
  A self-reported questionnaire that assesses manual ability in individuals with upper limb impairments. It consists of 23 items, where respondents rate the difficulty of performing daily activities using their hands. Scores are measured on a 3-point scale (0 = impossible, 1 = difficult, 2 = easy), with higher scores indicating better manual ability.
Change in Box and Blocks | Change from pre (week 3) to post intervention (week 8)
  An assessment of manual dexterity and upper limb function. It involves moving as many blocks as possible from one compartment of a box to another in 60 seconds using one hand. The score is based on the total number of blocks successfully transferred, with higher scores indicating better upper limb function.

OTHER OUTCOMES:
Demographic and stroke information questionnaire | baseline (week 0)
  To describe the participants
The Montreal Cognitive Assessment (MoCA) | Baseline (week 0)
  To describe the participants' cognitive status. Scores range between 0-30, a score of 26 or above is considered in the normal range.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Israel, Israel

IPD SHARING:
Plan to Share IPD: No